CLINICAL TRIAL: NCT02687100
Title: Does Beclomethasone Instillation Above the Cuff of Endotracheal Tubes Decrease the Occurrence of Postoperative Sore Throat? A Randomized Controlled Trial
Brief Title: The Effects of Beclomethasone Upper the Endotracheal Cuff on the Occurrence of Sore Throat at Extubation
Acronym: BEnTS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to instillation site of the cortisone and the development of the related SARS-Cov2 infection, it was preferred to terminate the trial and develop it again without beclomethasone
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Temistocle Taccheri, MD, resident of Department of Anesthesia and Intensive Care , Policlinico A. Gemelli , Catholic University of the Sacred Heart in Rome, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DMC
Record Dates: First submitted 2016-02-10; First posted 2016-02-22 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia, Endotracheal
Keywords: intubation; intensive care; cardiac surgery; sore throat
MeSH Terms: conditions — Pharyngitis | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beclomethasone (Experimental): Patients will receive beclomethasone, 0.8 mg of saline to a volume of 8 mL, three times through the line for suctioning above the cuff: a) after positioning the tube; b) at the arrival in the cardiac intensive care unit; c) just prior to start respiratory weaning. The solution will be aspirated 15 minutes after the instillation.
  Interventions: Drug: Beclomethasone
- Placebo (Placebo Comparator): Patients will receive 8 mL of saline without any drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beclomethasone — beclometasone, 0.8 mg of saline to a volume of 8 mL, three times through the line for suctioning above the cuff: a) after positioning the tube; b) at the arrival in the cardiac intensive care unit; c) just prior to start respiratory weaning
  Other Names: Qvar, Beclovent, Vanceril, Vanceril DS
  Arms: Beclomethasone
Drug: Placebo — patients will receive 8 mL of saline without any drug
  Arms: Placebo

SUMMARY:
The aim of the study is to test the effectiveness of a solutions of beclomethasone repeatedly instilled through the supraglottic line of the endotracheal tube on post-extubation airway disturbances related to tracheal intubation. The primary endpoint will be the decrease of the incidence of sore-throat 15 minutes and 12 hours after extubation. Secondary endpoints will regard the effects on hoarseness and cough.

DETAILED DESCRIPTION:
The study will be prospective, randomized, controlled. Patients will be premedicated with diazepam, 0.1 mg/Kg and scopolamine, 0.05 mg/Kg, i.m. one hour prior to their arrival in the operatory theatre. Anesthesia will be induced by fentanyl, 0.1 mg, and propofol, 1.5-2 mg/Kg. After obtaining muscle relaxation with cis-atracurium, 0.15 mg/Kg, a Taper Guard Evac Murphy Eye Oral Tracheal Tube (Mallinkrodt, Mirandola, Italy) with an internal diameter of 9 in men and 8 in women, will be positioned. These tubes have a line for suctioning above the cuff. The cuff pressure will be set to 20-30 cmH2O and checked every 6 hours with a proper inflating device. Patients will be connected to a mechanical ventilator and anesthesia will be maintained with sevoflurane 1-2.5% and remifentanil, 0.05-0.15 mcg/Kg/min. At the end of surgery, patients will be moved to the cardiac surgical intensive care, connected to a mechanical ventilator, and sedated with propofol and remifentanil until the conditions needed for weaning from the ventilator (control of bleeding, cardiovascular stability, thermal equilibrium) are achieved. Then, propofol infusion will be stopped and remifentanil dosage decreased to 0.02-0.05 mcg/Kg/min. After a successful t-tube trial of spontaneous breathing, tracheal tubes will be removed. Remifentanil infusion will be continued and dosage titrated on patient pain evaluated with a VAS scale; paracetamol 1 g will be given if need be.

ELIGIBILITY:
Inclusion Criteria:

* intensive care postoperative admission
* tracheal intubation for a total lapse of time between 10 and 18 hours

Exclusion Criteria:

* age < 18,
* hypersensitivity to FANS and/or corticosteroids,
* a medical history positive for diseases affecting upper airways or trachea or causing cough, hoarseness, or voice disorders;
* intubation after more than two attempts or with aids (i.e. stylets, Airtraq, Glidescope, Fibroscopy).

Ages: 18 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Decrease of the incidence of sore-throat. | Fifteen minutes after removing the tracheal tube
  Presence and intensity of sore throat by asking the patients to quantify it on a 0-3 scale
  Sore Throat Scoring System*
  0 No sore throat
  1. Minimal sore throat, less severe than with a cold
  2. Moderate sore throat, similar to that noted with a cold
  3. Severe sore throat, more severe than noted with a cold

SECONDARY OUTCOMES:
Decrease of the incidence of hoarseness | Fifteen minutes after removing the tracheal tube
  Presence and degree of hoarseness by asking the patients to quantify it on a 0-3 scale (table 3). In addition patients will be asked to pronounce a prolonged "e" in order to assess the capacity to adduce vocal cords, an ENT evaluation will be requested.
  Hoarseness Scoring System*
  0 No evidence of hoarseness
  1. Hoarseness that is noted by the patient only
  2. Hoarseness that is easily noted

CONTACTS AND LOCATIONS:
Overall Officials: Franco Cavaliere, MD, Principal Investigator — Department cardiovascular diseases A. Gemelli Polyclinic , University Sacred Heart in Rome

IPD SHARING:
Plan to Share IPD: Yes